CLINICAL TRIAL: NCT05120401
Title: Causal Relationship Between Dry Eye and Accommodative Spasm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Chin Mai, doctor, Far Eastern Memorial Hospital
Other Study IDs: 110100-E
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- dry eye with presbyopia: dry eye with presbyopia , Intervention : glasses prescrubed
  Interventions: Device: presbyopia glasses
- dry eye with presbyopia without glasses use: no glasses use
  Interventions: Device: presbyopia glasses

INTERVENTIONS:
Device: presbyopia glasses — fogging for glasses for far and intermediate

SUMMARY:
To investigate the causal relationship of Sicca dry eye patients with presbyopic refractive error and accommodative spasm.

DETAILED DESCRIPTION:
Dry eye is a disease of the ocular surface. Severe dry eye produce symptom of discomfort in and around the eye that drastically affect life quality of the patient. OSDI index is retrieve from a questionnaire specific for these dry eye symptoms, it is an internationally accepted level to reveal the severity of Dry eye disease. One part of the symptom is pain and soreness around the eye. Hyperalgesia is an increase response to a stressful/ noxious stimulus whereas allodynia is a painful response to a normally innocuous stimulus. Our hypothesis state that Sicca Dry eye upregulated inflammatory cytokine in the eye has pre-sensitized the nociceptor nerve fiber in the cornea and orbit, therefore the normally innocuous effort of accommodation and ciliary muscle contraction produce intolerable retro-orbital eye pain, which drives the patient to seek medical attention, on presentations these patient show an elevated OSDI and Pain Index (PI).

ELIGIBILITY:
Inclusion Criteria:

- dry eye

Exclusion Criteria:

* under 20 year old

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asian population with dry eye
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-11-05 (Estimated); Primary Completion 2024-07-20 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Improve of dry eye / OSDI | 30 days
  OSDI improve

CONTACTS AND LOCATIONS:
Overall Officials: Elsa LC MAI, MPH, Dr., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No